CLINICAL TRIAL: NCT07167498
Title: Continuous Remote Vital Sign Monitoring During Labour Analgesia With Remifentanil - a Prospective Observational Study
Brief Title: Continuous Remote Vital Sign Monitoring During Labour Analgesia With Remifentanil
Status: Not yet recruiting | Type: Observational
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Principal Investigator, Patricia Duch, Consultant, MD, Nordsjaellands Hospital
Other Study IDs: 104
Record Dates: First submitted 2025-09-02; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Labor Pain
Keywords: remifentanil; labour analgesia; remote monitoring; safety
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: The midwife stays in the labour room during remifentanil PCA for labour analgesia: Group 1: The midwife stays in the labour room while the parturient are having remifentanil for labour analgesia.
  Interventions: Behavioral: Intermittent midwife absence during remote monitoring of remifentanil PCA in labour
- Group 2: The midwife can leave the labour room during remifentanil PCA for labour analgesia: Group 2: the midwife is permitted to leave the labour room for intervals of up to 10 minutes while carrying a personal handheld device that displays continuous SpO₂, respiratory rate, and heart rate for remote monitoring.
  Interventions: Behavioral: Intermittent midwife absence during remote monitoring of remifentanil PCA in labour

INTERVENTIONS:
Behavioral: Intermittent midwife absence during remote monitoring of remifentanil PCA in labour — Midwife absence during remifentanil PCA for labour analgesia.
  We aim to include a total of 80 participants. All will receive remifentanil PCA for labour analgesia and be monitored with remote monitoring equipment. First a group of 40 parturients will be included, and the attending midwife will not be allowed to leave the parturient (Group 1). A following group of 40 parturients will then be included and the attending midwife can leave the room in intervals up to 10 minutes (Group 2).

SUMMARY:
Continuous remote vital sign monitoring during labour analgesia with remifentanil - a prospective observational study

Remifentanil PCA represents a well-tolerated, effective and valuable option for labour analgesia, yet its wider implementation is still limited by concerns of opioid side-effects particularly the risk of respiratory depression leading to desaturation, potentially affecting the foetus. Thus, continuous one-to-one observation and monitoring in the delivery room, with the midwife unable to leave the patient unattended, is recommended. Such constant one-to-one monitoring may be challenging in present health-care settings where staffing constraints may limit the implementation of remifentanil as routine obstetric care.

Continuous remote vital sign monitoring to display oxygen saturation (SpO₂), respiratory rate, and heart rate on a handheld device (smartphone), has the potential to address this barrier by allowing the midwife to leave the labour room for short, predefined intervals while maintaining continuous surveillance of maternal vital signs. Such an approach could free staff resources without compromising patient safety. While centralised foetal monitoring (CTG) is standard practice in many units, the application of continuous remote vital sign monitoring for women receiving remifentanil during labour has, to our knowledge, never been formally studied.

Objectives The aim is to study whether remote monitoring during remifentanil patient-controlled analgesia (PCA) for labour affects the incidence of maternal desaturation and other safety outcomes (bradypnoea, bradycardia, and neonatal outcomes, assessed via Apgar scores and umbilical cord pH.) The study will be conducted in a setting where remifentanil PCA is administered for labour analgesia and the midwife is permitted to leave the labour room for intervals of up to 10 minutes while the woman is remotely monitored using a handheld device carried by the midwife. Predefined criteria for when the woman must be accompanied (e.g., if SpO₂ < 94%, supplemental oxygen >2L/min., or decreased consciousness). Outcomes in this group will be compared with a control group where the midwife remains continuously present in the labour room.

DETAILED DESCRIPTION:
Introduction Remifentanil, a potent, ultra-short-acting opioid, administered intravenously via patient-controlled analgesia (PCA) has been used for more than a decade in several countries, particularly in Switzerland and at the Ulster Hospital in Ireland. In 2024, remifentanil was formally included as a standard option for labour analgesia in the United Kingdom and incorporated into the guidelines from the National Institute for Health and Care Excellence (NICE). The REMIPCA SAFE Network collaboration has further demonstrated that remifentanil PCA is a safe and effective method for labour analgesia, offering rapid onset, patient autonomy, and high maternal satisfaction (remiPCA.org).

In many European and Anglophone countries, nitrous oxide and epidural analgesia remain the most commonly used pharmacological methods for labour analgesia, while the use of remifentanil is not yet widespread in all settings. Nitrous oxide cause nausea and is under increasing scrutiny due to environmental concerns, while epidural analgesia, although highly effective for pain relief, is more invasive, resource intensive and associated with rare but severe complications.

Remifentanil PCA represents a well-tolerated, effective and valuable option for labour analgesia, yet its wider implementation is still limited by concerns of opioid side-effects particularly the risk of respiratory depression leading to desaturation, potentially affecting the foetus. Thus, continuous one-to-one observation and monitoring in the delivery room, with the midwife unable to leave the patient unattended, is recommended. Such constant one-to-one monitoring may be challenging in present health-care settings where staffing constraints may limit the implementation of remifentanil as routine obstetric care.

Continuous remote vital sign monitoring to display oxygen saturation (SpO₂), respiratory rate, and heart rate on a handheld device (smartphone), has the potential to address this barrier by allowing the midwife to leave the labour room for short, predefined intervals while maintaining continuous surveillance of maternal vital signs. Such an approach could free staff resources without compromising patient safety. While centralised foetal monitoring (CTG) is standard practice in many units, the application of continuous remote vital sign monitoring for women receiving remifentanil during labour has, to our knowledge, never been formally studied.

Objectives The aim is to study whether remote monitoring during remifentanil for labour analgesia affects the incidence of maternal desaturation and other safety outcomes (bradypnoea, bradycardia, and neonatal outcomes, assessed via Apgar scores and umbilical cord pH.) This will be assessed in a setup where remifentanil PCA for labour analgesia is given and the midwife is allowed maximum absence intervals of 10 minutes with predefined criteria for when the woman must be accompanied (e.g., if SpO₂ < 94%, supplemental oxygen >2L/min., or decreased consciousness) and compared with a control group where the midwife is in the labour room continuously.

Methods

Ethics The study will be conducted in compliance with the Declaration of Helsinki. Participation will be voluntary, and written informed consent will be obtained prior to inclusion. Participants may withdraw their consent at any time without consequences for their further treatment. Approval for data collection, processing, and storage will be sought from the Data Protection Authority for the Capital Region of Denmark prior to study initiation. The National committee on health research ethics, Denmark has approved the study in accordance with Danish legislation (ID: 2203648, date: 2024-06-25). All collected data will be handled in strict confidence and anonymised prior to analysis. The study protocol will be registered at ClinicalTrials.gov before inclusion of the first patient.

Study design A single centre before and after prospective observational study. Based on maternal and neonatal physiological parameters in parturients giving birth with remifentanil PCA for labour analgesia, using continuous remote vital sign monitoring, while the attending midwife is either continuously present in the labour room (group 1) or intermittently present, with absence intervals of up to 10 minutes (group 2)

Setting Location The study will be conducted at the labour ward of North Zealand Hospital. Recruitment period Recruitment is expected to be completed between 1 October 2025 and 31 December 2026.

Data collection Continuous monitoring of oxygen saturation (SpO₂), cardiotocography (CTG), respiratory rate, and heart rate during labour will be registered for analysis. Oxygen saturation (SpO₂), respiratory rate, and heart rate will be collected using the WARD technology (WARD247 Aps, Copenhagen, Denmark) and consists of threadless body-sensors which monitor oxygen saturation (SpO₂), ECG and respiratory rate every minute. These data are then electronically transferred to the WARD monitoring application on a handheld mobile device (smartphone). The adhesive body sensors are applied using a bracelet for the wrist and two ECG electrodes on the chest allowing considerable freedom of movement. CTG will be collected with Umbilical cord pH will be measured in all participants. Additional maternal and neonatal physiological parameters will be obtained from health records from the birth admission. The midwife will register when they are absent from the labour room, including frequency and duration of absences.

Remifentanil administration for labour analgesia Remifentanil is administered as patient-controlled analgesia (PCA) via an intravenous line. When the parturient presses the PCA button, a bolus of 20 µg remifentanil (corresponding to 1 mL) is delivered; the bolus dose may be adjusted between 10 µg and 30 µg. The lockout interval is 2 minutes. Administration must be discontinued around 10 minutes prior to delivery. The parturient is monitored for oxygen saturation (SpO₂), respiratory rate, cardiotocography (CTG), and heart rate. Each parturient will receive one-to-one midwifery care, as is standard practice in Denmark. The use of labour analgesia will be adapted to the individual course of labour, and medical pain management during active labour may include nitrous oxide, remifentanil, and epidural analgesia.

In the department's standard operating procedure, adapted from remipca.org, the target oxygen saturation (SpO₂) during the use of remifentanil is > 93%. If SpO₂ is < 94% for more than two minutes supplemental oxygen should be administered, either via face mask for short desaturation episodes or via nasal cannula.

When the parturients are receiving remifentanil for labour analgesia in the study protokol:

Group 1: The midwife stays in the labour room Group 2: the midwife is permitted to leave the labour room for intervals of up to 10 minutes while carrying a personal handheld device that displays continuous SpO₂, respiratory rate, and heart rate for remote monitoring. The monitoring system presents SpO₂, HR and RR continuously on the screen (updated every minute), and the midwife is responsible for continuous observation via the remote monitoring system and must respond immediately if SpO₂ falls below 94% or RR are below 10. As a safety precaution, an alarm is triggered after 10 minutes if SpO2 falls below 88%, after 5 minutes if SpO₂ falls below 85%, and immediately if SpO₂ falls below 80% and immediately if RR falls to ≤5 brpm.

The midwife is only permitted to leave the labour room if the parturient receiving remifentanil is awake, responsive, and accompanied by a partner who is capable and instructed to call for assistance if SpO₂ drops below 94% or if the parturient becomes unconscious. CTG will be centrally monitored at the ward level by the ward responsible midwife, who maintains an overview of CTG tracings from all delivery rooms.

As an extra safety precaution during this study, the ward-responsible midwife will also be informed if the attending midwife leaves the room and will be able to monitor the SpO₂ together with the CTG via the central monitoring system connected to all delivery rooms.

ELIGIBILITY:
Inclusion criteria:

* Minimum 18 years of age
* Able to provide written informed consent
* Giving birth to a singleton, cephalic presenting, expected healthy child, gestational age > 37 weeks.
* In active labour

Exclusion criteria

* Respiratory or cardiac disease
* BMI ≥ 40 Other opioids within the last 4 hours.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will be conducted at the labour ward of North Zealand Hospital. All parturients who meet the eligibility criteria may be included, provided that qualified staff are available at the time of admission.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of SpO₂ 90-93% lasting more than 2 minutes | During labour
  During the use of remifentanil for labour analgesia.

SECONDARY OUTCOMES:
Incidence of SpO2 89-85% lasting more than one minute | During labour
  During the use of remifentanil for labour analgesia.
Any incidence of SpO2 < 85% | During labour
  During the use of remifentanil for labour analgesia.
Incidence of RR < 9 for ≥5 minutes | During labour
  During the use of remifentanil for labour analgesia.
Incidence of neonates with Apgar score < 7 | measured 5 minutes after birth
  During the use of remifentanil for labour analgesia.

OTHER OUTCOMES:
Incidence of parturient being unconscious assessed by AVPU assessment scale (Alert, Voice, Pain, Unresponsive) during the use of remifentanil for labour analgesia. | During the use of remifentanil for labour analgesia.
  During the use of remifentanil for labour analgesia.
Incidence of HR < 50 | During the use of remifentanil for labour analgesia.
  During the use of remifentanil for labour analgesia.
Incidence of RR ≤5 | During the use of remifentanil for labour analgesia.
  During the use of remifentanil for labour analgesia.
Incidence of neonates with umbilical cord pH < 7.00 | measured within minutes after birth
  During the use of remifentanil for labour analgesia.
Cumulative duration of SpO2 <85% per patient | During labour
  During the use of remifentanil for labour analgesia.
Cumulative duration SpO2 89-85% per patient | During labour
  During the use of remifentanil for labour analgesia.
Cumulative duration of SpO2 90-94% per patient | During labour
  During the use of remifentanil for labour analgesia.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Duch, MD, Principal Investigator — Nordsjaellands Hospital
Locations (1):
- University Hospital of Copenhagen, Northern Zealand, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: No